CLINICAL TRIAL: NCT07244926
Title: Sacituzumab Tirumotecan (Sac-TMT) Plus Bevacizumab in Second-line Treatment of Advanced Non-squamous Non-small Cell Lung Cancer (NSCLC) Without Actionable Gene Alterations: a Single-arm, Phase II Trial
Brief Title: Sac-TMT Plus Bevacizumab as Second-Line Treatment for Advanced Non-Squamous Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-IIT-019
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sac-TMT plus bevacizumab (Experimental)
  Interventions: Drug: Sacituzumab tirumotecan plus bevacizumab

INTERVENTIONS:
Drug: Sacituzumab tirumotecan plus bevacizumab — The eligible patients will receive intravenous sac-TMT 4mg/kg every 2 weeks plus intravenous bevacizumab 10mg/kg every 2 weeks until disease progression, death, unacceptable toxicity, or another treatment discontinuation criterion is met.

SUMMARY:
In this single-arm, phase II study, we aimed to evaluate the efficacy and safety of sac-TMT plus bevacizumab in patients with advanced non-squamous NSCLC who showed disease progression on or after first-line ICI plus platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old, regardless of gender
* Histologically or cytologically confirmed locally advanced or metastatic non-squamous NSCLC (stage IIIB/C or IV not amenable to curative treatment)
* Negative for EGFR sensitizing mutations [no exon 19 deletion (19-Del) or exon 21 point mutation (L858R mutation)] and ALK fusion gene, and no known actionable gene alterations in ROS1, NTRK, BRAF, MET, KRAS, HER2, or RET.
* Disease progression after first-line platinum-based chemotherapy combined with anti-PD-(L)1 therapy.
* At least one measurable lesion according to RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 within 7 days prior to administration.
* Expected life expectancy ≥ 12 weeks.
* Adequate organ and bone marrow function.
* Agreement to use effective medical contraception methods from the time of signing the informed consent form until 6 months after the last dose for female subjects of childbearing potential and male subjects with partners of childbearing potential.
* Join the study voluntarily, signs the informed consent form, and is able to comply with the visits and related procedures stipulated in the protocol.

Exclusion Criteria:

* Histologically or cytologically confirmed squamous cell NSCLC or mixed with small cell lung cancer, neuroendocrine carcinoma, or carcinosarcoma components.
* Previously received any of the following treatments (including in the adjuvant or neoadjuvant setting): a) Therapy targeting TROP2. b) Any drug therapy containing a topoisomerase I inhibitor, including Antibody-Drug Conjugate (ADC) therapy. c) Anti-angiogenic agents.
* Requirement for strong inhibitors or inducers of Cytochrome P450 3A4 (CYP3A4) within 2 weeks prior to the first dose or during the study period.
* Documented severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or history of corneal disease that prevents/delays corneal healing.
* Known leptomeningeal metastasis, brainstem metastasis, spinal cord metastasis and/or compression, or active central nervous system (CNS) metastases. Subjects with brain metastases previously treated with local therapy can participate if they are clinically stable for at least 4 weeks prior to dosing and do not require corticosteroids or anticonvulsants for at least 14 days; subjects with untreated asymptomatic brain metastases may be enrolled after investigator assessment.
* History of other malignancies within 3 years prior to dosing (except for tumors cured with local therapy, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, etc.).
* Presence of severe cardiovascular or cerebrovascular diseases or risk factors.
* Uncontrolled systemic diseases, as judged by the investigator.
* Urinalysis shows urine protein ≥ ++ and confirmed 24-hour urine protein quantification > 1.0 g.
* History of (non-infectious) interstitial lung disease (ILD) or non-infectious pneumonitis requiring steroid treatment, current ILD or non-infectious pneumonitis, or suspected ILD or non-infectious pneumonitis that cannot be ruled out by imaging at screening.
* Clinically severe pulmonary impairment due to concurrent pulmonary diseases.
* Subjects with active chronic inflammatory bowel disease, gastrointestinal obstruction, severe ulcer, gastrointestinal perforation, intra-abdominal abscess, or acute gastrointestinal bleeding.
* Tumor invasion or compression of surrounding vital organs and blood vessels accompanied by related symptoms (e.g., superior vena cava syndrome), or risk of esophagotracheal fistula or esophagopleural fistula.
* History of bleeding tendency or coagulation disorder and/or clinically significant bleeding symptoms or risks within 4 weeks prior to the first dose.
* Use of aspirin (>325 mg/day) or treatment with dipyridamole or clopidogrel within 2 weeks prior to the first dose.
* Use of full-dose oral or intravenous anticoagulants or thrombolytic agents within 2 weeks prior to the first dose.
* Biopsy or other minor surgery (excluding placement of vascular access devices) within 7 days prior to the first dose.
* Toxicity from previous anti-tumor therapy has not recovered to ≤ Grade 1 or the level specified in the eligibility criteria (except for toxicities judged by the investigator to pose low safety risks, such as alopecia, fatigue, etc.).
* Known active tuberculosis. Subjects suspected of having active tuberculosis require clinical evaluation to exclude it.
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Active Hepatitis B or Hepatitis C. Note: Subjects who are HBsAg positive are required to receive anti-hepatitis B virus therapy during the study treatment period.
* Positive human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
* Known allergy to the investigational drug or any of its components, history of severe hypersensitivity reactions to other biological agents.
* Major surgery within 4 weeks prior to dosing or anticipated need for major surgery during the study period.
* Severe infection within 4 weeks prior to dosing, active infection requiring systemic anti-infective therapy within 2 weeks prior to dosing.
* Non-specific immunomodulatory therapy within 2 weeks prior to dosing.
* Radiation therapy to lung lesions with a total dose > 30 Gy within 6 months prior to dosing; non-thoracic radiotherapy with a total dose > 30 Gy or extensive radiotherapy (including radionuclide therapy such as Strontium-89) within 4 weeks prior to dosing; palliative radiotherapy for symptom control is allowed but must be completed at least 2 weeks before the first dose.
* Administration of live vaccines within 30 days prior to dosing, or planned administration of live vaccines during the study period.
* Rapid deterioration of condition during the screening period prior to dosing.
* Pregnant or lactating women.
* Local or systemic diseases caused by non-malignant conditions, or diseases or symptoms secondary to the tumor, that could lead to high medical risk and/or uncertainty in survival assessment.
* Any condition that, in the investigator's judgment, interferes with the evaluation of the investigational product, subject safety, or interpretation of study results, or any other situation where the investigator considers the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to approximately 60 months
  ORR is defined as the proportion of patients with a confirmed complete (CR) or partial response (PR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Disease control response (DCR) | up to approximately 60 months
  DCR is defined as the proportion of patients with the best overall response of CR, PR, and stable disease (SD) Per RECIST 1.1 as assessed by the investigator.
Duration of response (DOR) | Until progression or death, up to approximately 60 months
  DOR is defined as first documented evidence of a CR or PR until PD or death
Progression-free survival (PFS) | Until progression or death, up to approximately 60 months
  PFS is defined as the time from the initial treatment to the first occurrence of disease progression or death (whichever occurs first)
Overall Survival (OS) | Until death, up to approximately 60 months.
  OS is defined as the time from the initial treatment to the date of death due to any cause.
Incidence and severity of adverse events (AEs) | up to approximately 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiubao Ren, MD. Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Liang Liu, MD. Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China